CLINICAL TRIAL: NCT03229681
Title: Baduanjin Exercise for Patients With Chronic Heart Failure on Phase II Cardiac Rehabilitation: A Prospective, Randomized, Controlled Clinical Trial
Brief Title: Baduanjin Exercise for Patients With Chronic Heart Failure on Phase II Cardiac Rehabilitation
Acronym: BEPCR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20170506
Record Dates: First submitted 2017-07-23; First posted 2017-07-25 (Actual); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Rehabilitation With CHF; NYHA Class I or II
Keywords: Baduanjin; CHF; 6MWT; CPET
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baduanjin exercise group (Experimental): Participants in this group received routine rehabilitation training and Baduanjin exercise
  Interventions: Behavioral: Baduanjin exercise
- Routine rehabilitation group (Active Comparator): Participants in this group only received routine rehabilitation training
  Interventions: Behavioral: Routine rehabilitation group

INTERVENTIONS:
Behavioral: Baduanjin exercise — Participants in this groups received routine rehabilitation training and Baduanjin exercise. During the period of rehabilitation, physicians provides a wide range of medical, nutrition and mental health counseling, as well as rational drug-treatment. Baduanjin exercise protocol according to the "Health Qigong Baduanjin Standard" enacted by the General Administration of Sports in 2003. Due to the low-activity tolerance of CHF patients, we performed with a refined version of Baduanjin. Each Baduanjin exercise session lasts 45 minutes and continues twice per week for 12 weeks.
  Other Names: Routine rehabilitation
  Arms: Baduanjin exercise group
Behavioral: Routine rehabilitation group — Participants in this qroup only received the routine rehabilitation training. During the period of rehabilitation, physicians provides a wide range of medical, nutrition and mental health counseling, as well as rational drug-treatment. They should also come to rehabilitation center for physical exercise,45 minutes per day，twice per week, lasts 12 weeks.
  Arms: Routine rehabilitation group

SUMMARY:
Chronic heart failure (CHF) is the end stage of various kinds of cardiovascular diseases with high mortality. After a long period of medical treatment or surgical treatment, patients suffered great pain physically and mentally. How to improve the quality of life and prognosis in patients with CHF, which is a hot topic in the field of cardiac rehabilitation now. Baduanjin, as one of the traditional Chinese qigong exercises, has the features of generous stretch, soft consistency, dynamic but static, which is an appropriate movement pattern for CHF patients.

To investigate the efficacy and safety of Baduanjin exercise for patients with coronary heart disease complicated with chronic heart failure (CHF). A randomized, controlled and prospective clinical trial was designed.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 40 to 75 years;
* Diagnosed with chronic heart failure caused by coronary heart disease;
* NYHA class I or II;
* Patients with an ejection fraction (LVEF) more than 40%;
* Participants in accordance with the guidelines define as stage II cardiac rehabilitation;
* Participants signed the informed consent freely and voluntarily.

Exclusion Criteria:

* The condition was serious or movement restrained by other diseases;
* In the acute stage of chronic heart failure;
* Participants with poorly control of blood pressure (SBP≥180mmHg or DBP≥100mmHg);
* Resting heart rate is beating over 120 beats a minute, or merged with malignant arrhythmia;
* Participants who have contraindications to cardiopulmonary test or exercise training;
* Patients who have other serious acute， chronic organic disease or mental disorders;
* Participants practiced in any kinds of traditional Chinese medicine exercises in last three months.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-05-02 (Actual); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Six-minute walk test（6MWT） | Baseline, 3 months
  Testing patients changes on walking distance and accompanies symptoms in 6 minutes

SECONDARY OUTCOMES:
Cardiopulmonary exercise test (CPET) | Baseline, 3 months
  CPET including peak VO2 (ml/kg/min)， AT，VE/VCO2, et,al.
Left ventricular ejection fraction（LVEF） | Baseline, 3 months
Left ventricular end-diastolic diameter (LVDD) | Baseline, 3 months
Minnesota living with heart failure questionnaire (MLHFQ) | Baseline, 3 months
  Record the quality of life of patients with heart failure
NT-proBNP | Baseline, 3 months
hs-CRP | Baseline, 3 months
HRV | Baseline, 3 months
  Mainly includes SDANN Index, SDNN Index
Major adverse cardiovascular events (MACE) | Baseline, 3 months, 6months
  Defined as death, myocardial infarction (MI), stroke and re-hospitalization related to cardiovascular disease
NYHA classification | Baseline, 3 months, 6months
  The changes of heart function were compared after treatment
The Main TCM symptoms | Baseline, 3 months
  The changes of scores of TCM syndromes

CONTACTS AND LOCATIONS:
Overall Officials: Hao Xu, Study Director — Xiyuan Hospital of China Academy of Chinese Medical Sciences
Locations (1):
- Xiyuan Hospital of China Academy of Chinese Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yu M, Li S, Li S, Li J, Xu H, Chen K. Baduanjin exercise for patients with ischemic heart failure on phase-II cardiac rehabilitation (BEAR trial): study protocol for a prospective randomized controlled trial. Trials. 2018 Jul 16;19(1):381. doi: 10.1186/s13063-018-2759-4. PMID 30012193